CLINICAL TRIAL: NCT05583500
Title: Phase Angle as a Marker of Muscle Damage, Muscle Fatigue and Inflammation, After Eccentric Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UFV-JB22
Record Dates: First submitted 2022-09-29; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Phase Angle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group: excentric exercise protocol (Experimental): Excentric exercise protocol will be performed for all subjets, consisted of 10 sets of 20 repetitions of squats, jumping from a height of 50 cm
  Interventions: Other: Experimental: Single group: excentric exercise protocol

INTERVENTIONS:
Other: Experimental: Single group: excentric exercise protocol — Excentric exercise protocol will be performed for all subjets, consisted of 10 sets of 20 repetitions of squats, jumping from a height of 50 cm

SUMMARY:
The purpose of this study will be to assess the effectiveness of bioimpedance device (BIA) as a safe, rapid, and non-invasive method of analyzing muscle damage induced by high intensity induced eccentric exercise as an alternative measurement tool against traditional assessment methods.

A sample of 28 sedentary subjects will be recruited, all participants will perform an eccentric exercise protocol.

Measurements will be done before performing the exercise protocol, immediately after finishing the protocol, 3h after the end of the exercise protocol, 24h after the end of the exercise protocol and 48h after the end of the exercise protocol.

The variables analyzed in all subjects will be phase angle, creatinkinase, jumping strength, VAS scale, white blood count cell, quadriceps muscle thickness, Borg scale and anxiety and depression questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjets
* Sedentary subjects

Exclusion Criteria:

* Trained subjects
* Subjects with musculoskeletal pathology
* Previous Surgeries in the last 6 months
* Subjects under pharmacological treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Phase angle | change from baseline to 72 hours
  The phase angle, which is measured via bioelectrical impedance analysis (BIA), InBody 770 ,is a clinically important bioimpedance parameter used for nutritional assessment and evaluating the risk of various diseases. The phase angle was calculated automatically by the BIA device from these two components according to the following formula: phase angle (°) = (reactance/resistance) × (180°/π).

SECONDARY OUTCOMES:
Pain: VAS | change from baseline to 72 hours
  Visual Analogic Scale. Pain will be measured with a visual analog scale from 0 to 10. 0 points is no pain.
Quadriceps thickness | change from baseline to 72 hours
  Quadriceps muscle thickness will be measures in mm. by an ultrasound device
Creatinkinase (CK concentration) | change from baseline to 72 hours
  CK concentration will be measure in mg/dl with a portal analyzer (SpotchemTM EZ SP-4430), using test strips.
cellular inflammatory markers | change from baseline to 72 hours
  Cellular inflammatory markers will be measured with hematology analyzer (Sysmex KX-21N Automed) in 10^9/L and % White blood count, lymphocytes, neutrophils, monocytes, eosinophils, basophils will be analyzed
Leg power | change from baseline to 72 hours
  Leg power will be assessed using vertical jump test, with Chronojump platform (CHRONOJUMP Boscosystem)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Buffet García, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No